CLINICAL TRIAL: NCT06441032
Title: Survival of Cast Restorations - Restorations Made of Precious Metal vs. Non-precious Metal
Brief Title: Retrospective Database Study: Survival of Cast Restorations - Restorations Made of Precious Metal vs. Non-precious Metal
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, PD Dr. med. dent., Dr. rer. medic., Senior Lecturer, University Medical Center Goettingen
Other Study IDs: Survival-Cast-Restorations; 21/11/22 (Other: Local Ethics Commission)
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Dental Restoration Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Precious metal: Single-tooth cast restorations made of precious metal.
  Interventions: Other: No patient treatment is associated with the study
- Non-precious metal: Single-tooth cast restorations made of non-precious metal
  Interventions: Other: No patient treatment is associated with the study

INTERVENTIONS:
Other: No patient treatment is associated with the study — No patient treatment is associated with the study.

SUMMARY:
The aim of this study is to determine and compare the longevity of single-tooth cast restorations made of precious metal vs. non-precious metal (e.g. partial crowns, crowns) and to determine the influence of patient-, tooth-, treatment-, and restoration-specific parameters on longevity.

Patients who received single-tooth cast restorations made of precious metal or non-precious metal (e.g. partial crowns, crowns) between 1997 and 2022 will be retrospectively analyzed. Patient-, tooth-, treatment-, and restoration-specific parameters will be obtained from digital and paper-based dental records.

Survival and success of the restorations will be assessed using Kaplan-Meier statistics. Mean annual failure rates (mAFR) and median survival time will be calculated (Kaplan-Meier statistics). Potential predictive factors will be tested using log-rank tests and multi-variate Cox-regression analysis.

DETAILED DESCRIPTION:
No patient treatment is associated with the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients insured in the statutory health insurance.
* Patients who received single-tooth cast restorations made of precious metal or non-precious metal (e.g. partial crowns, crowns) within the Department of Preventive Dentistry, Periodontology and Cariology between 1997 and 2022.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients insured in the statutory health insurance who received single-tooth cast restorations made of precious metal or non-precious metal (e.g. partial crowns, crowns) within the Department of Preventive Dentistry, Periodontology and Cariology between 1997 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Success of restoration | 1997-2023
  Success is defined as the time-interval without a subsequent re-intervention of the restoration or extraction of the tooth.

SECONDARY OUTCOMES:
Survival of restoration | 1997-2023
  Survival is defined as the time-interval without replacement of the restoration or extraction of the tooth.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No